CLINICAL TRIAL: NCT02251457
Title: Open Label Trial of Ranolazine in Myotonia Congenita, Paramyotonia Congenita, & Myotonic Dystrophy Type 1
Brief Title: Study of Ranolazine in Myotonia Congenita, Paramyotonia Congenita and Myotonic Dystrophy Type 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, William Arnold, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-259-1605; IN-US-259-1605 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Myotonia Congenita; Paramyotonia Congenita; Myotonic Dystrophy 1
Keywords: Myotonia Congenita; ranolazine; Ohio State; Open Label; Paramyotonia Congenita; Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonia Congenita; Myotonic Disorders; Myotonic Dystrophy | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranolazine (Experimental): ranolazine 500mg, twice daily for two weeks; 1000mg twice daily for 2 weeks
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — Ranexa is FDA approved for chronic angina
  Other Names: Ranexa®

SUMMARY:
The purpose of this study is to gather preliminary data to determine if ranolazine is a safe and effective treatment for the symptoms of myotonia congenital, paramyotonia congenita, and myotonic dystrophy type 1. The duration of the study is 5 weeks.

DETAILED DESCRIPTION:
Recent advances in the understanding of myotonia congenita have identified potential areas that could possibly respond to treatment in a drug study. The drug ranolazine (trade name Ranexa) is a FDA-approved medication to treat chest pain in patients with heart disease. Ranolazine has been studied in mice with myotonia congenita. The data from this animal model suggest that ranolazine may improve the symptoms and signs of myotonia. All individuals that participate will be placed on active drug. The investigators want to see if this drug is safe to take without causing too many side effects for people with myotonia congenita, paramyotonia congenital and myotonic dystrophy type 1. Participants will go to The Ohio State University for study visits. Participants will take ranolazine for four weeks. Participants can expect a total of 4 study visits and 2 phone calls over the 5 week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myotonia congenital, paramyotonia congenital or Myotonic Dystrophy Type 1 established by genetic testing in the subject or in a first-degree relative.
* Clinically evident myotonia

Exclusion Criteria:

* Contraindications to ranolazine use:

  * for fungus infection: ketoconazole (Nizoral), itraconazole (Sporanox, Onmel)
  * for infection: clarithromycin (Biaxin)
  * for depression: nefazodone
  * for HIV: nelfinavir (Viracept), ritonavir (Norvir), lopinavir and ritonavir (Kaletra), indinavir (Crixivan), saquinavir (Invirase).
  * for tuberculosis (TB): rifampin (Rifadin), rifabutin (Mycobutin), rifapentine (Priftin)
  * for seizures: phenobarbital, phenytoin (Phenytek, Dilantin, Dilantin-125), carbamazepine (Tegretol)
  * the herbal supplement St. John's wort

    * you have scarring (cirrhosis) of your liver
* Concurrent use of mexiletine, lacosamide, acetazolamide, phenytoin, quinine, procainamide, Saint John wort or tocainide. Patients who were previously treated with these medications may participate. They need to be off of the medication for at least a week prior to enrollment.
* QTc >470 ms for men and >480 ms for women.
* Women who are pregnant or breastfeeding
* Direct family history of sudden cardiac death

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-08; Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Questionnaires: Short Form Health Survey (SF-36) and Individualized Neuromuscular Quality of Life Questionnaire (INQoL) | 1 month
  quality of life measurements for overall health and neuromuscular disease
Muscle tasks | 1 month
  The subject is observed and timed while rising from an arm chair, walking 3 meters, turning, walking back, and sitting down again
Electromyography (EMG) Myotonia | 1 month
  To see if the electrical potentials produced by the muscle fibers change.

SECONDARY OUTCOMES:
Electrocardiogram (ECG) | 1 month
  to measure heart function and observe QT interval (a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle)

CONTACTS AND LOCATIONS:
Overall Officials: William D Arnold, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Novak KR, Norman J, Mitchell JR, Pinter MJ, Rich MM. Sodium channel slow inactivation as a therapeutic target for myotonia congenita. Ann Neurol. 2015 Feb;77(2):320-32. doi: 10.1002/ana.24331. Epub 2015 Jan 9. PMID 25515836
- [Derived] Spillane J, Trip J, Drost G, Faber CG, Hanna MG, Nevitt SJ, Vivekanandam V. Drug treatment for myotonia. Cochrane Database Syst Rev. 2025 Apr 8;4(4):CD004762. doi: 10.1002/14651858.CD004762.pub3. PMID 40197813
- [Derived] Lorusso S, Kline D, Bartlett A, Freimer M, Agriesti J, Hawash AA, Rich MM, Kissel JT, David Arnold W. Open-label trial of ranolazine for the treatment of paramyotonia congenita. Muscle Nerve. 2019 Feb;59(2):240-243. doi: 10.1002/mus.26372. Epub 2018 Dec 21. PMID 30390395